CLINICAL TRIAL: NCT03887845
Title: A Prospective Case-control Study Comparing the Effects of Open and Laparoscopic Gastrointestinal Surgery on Gastrointestinal Function
Brief Title: Effects of Open and Laparoscopic Gastrointestinal Surgery on Gastrointestinal Function
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yong Zhou, Clinical Professor, West China Hospital
Other Study IDs: 858105185
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Postoperative Ileus
Keywords: postoperative ileus; prospective study; case-control; open surgery; laparoscopic surgery; bowel recovery; intestinal recovery; gut recovery
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open gastrointestinal surgery: All patients enrolled in this group would undergo open gastric and colorectal resection surgery.
  Interventions: Procedure: Surgery
- Laparoscopic gastrointestinal surgery: All patients enrolled in this group would undergo laparoscopic gastric and colorectal resection surgery.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — The respective surgical approach for any gastric and colorectal surgery

SUMMARY:
A prospective study to compare the postoperative ileus in open and laparoscopic gastrointestinal surgery through the determination of the time the patient takes to pass flatus, pass stool, bowel movement, oral intake, the time of hospital stay and total hospital costs. Postoperative ileus (POI) is one of the major focus of concern for surgeons, hospital executives, quality assurance directors as well as patients because of its role in causing patient distress, discomfort, and morbidity, leading to an increase in the duration of hospital stay and cost of care.

DETAILED DESCRIPTION:
All patients aged ≥18 years scheduled to undergo gastric and colorectal cancer resection surgery at the Department of Gastrointestinal Surgery, West China Hospital between 2019 to 2020 will be screened for eligibility. The inclusion criteria for the study will be the patient undergoing elective gastric cancer surgery, have the American Society of Anesthesiologist (ASA) grade ≤ III, alert consciousness, and BMI, and accurate preoperative diagnosis of gastric adenocarcinoma on the basis of computed tomography CT scan report, Gastroscopy and Histopathological reports. Exclusion criteria will be those who cannot participate in study assessments owing to the language barrier, dementia or postoperative delirium; previously received palliative surgery, develops early postoperative bowel obstruction, Anastomotic leakage or Gastroparesis, those requiring reoperation for any other indication before the commencement of formal assessment for PPOI. Those requiring more than 30 minutes of adhesiolysis. Each patient will be approached during preoperative counseling on an individual basis by one of the authors (YZ)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years scheduled to undergo elective abdominal surgery
* American Society of Anesthesiologist (ASA) grade ≤ III
* Alert consciousness
* Any BMI
* Accurate preoperative diagnosis on the basis of necessary reports

Exclusion Criteria:

* Cannot participate in study assessments owing to the language barrier, dementia or postoperative delirium
* Previously received palliative surgery
* Develops early postoperative bowel obstruction, Anastomotic leakage or Gastroparesis
* Those requiring reoperation for any other indication before the commencement of formal assessment for POI
* Those requiring more than 30 minutes of adhesiolysis
* Emergency cases
* American Society Anesthesia (ASA) class IV or V patients, pregnancy, patient with abdominal carcinomatosis or radiation enteritis, inoperable cases due to metastasis, patients simultaneously enrolled in any other competing for clinical study and violation of study protocol by the patient or patient care team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients enrolled in this study would undergo gastric and colorectal resection surgery
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Time to first flatus | up to 1-4 Days after surgery
  The time between end of surgery and passage of first flatus
Length of hospital stay | up to 1-10 Days after surgery
  The time between end of surgery and written discharge ticket

SECONDARY OUTCOMES:
Time to first bowel movement | up to 1-6 Days after surgery
  The time between end of surgery and first bowel movement
Time to first oral intake | up to 1-6 Days after surgery
  The time between end of surgery and first oral intake >25% than usual intake
Time to first defecation | up to 1-6 Days after surgery
  The time between end of surgery and first stool passage
Time to first ambulation | up to 1-6 Days after surgery
  The time between end of surgery and first time ambulation from bed

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cho JS, Kim HI, Lee KY, Son T, Bai SJ, Choi H, Yoo YC. Comparison of the effects of patient-controlled epidural and intravenous analgesia on postoperative bowel function after laparoscopic gastrectomy: a prospective randomized study. Surg Endosc. 2017 Nov;31(11):4688-4696. doi: 10.1007/s00464-017-5537-6. Epub 2017 Apr 7. PMID 28389801
- [Result] Gomez-Pinilla PJ, Binda MM, Lissens A, Di Giovangiulio M, van Bree SH, Nemethova A, Stakenborg N, Farro G, Bosmans G, Matteoli G, Deprest J, Boeckxstaens GE. Absence of intestinal inflammation and postoperative ileus in a mouse model of laparoscopic surgery. Neurogastroenterol Motil. 2014 Sep;26(9):1238-47. doi: 10.1111/nmo.12376. Epub 2014 Jun 26. PMID 24966010
- [Result] Yamamoto S, Hinoi T, Niitsu H, Okajima M, Ide Y, Murata K, Akamoto S, Kanazawa A, Nakanishi M, Naitoh T, Kanehira E, Shimamura T, Suzuka I, Fukunaga Y, Yamaguchi T, Watanabe M; Japan Society of Laparoscopic Colorectal Surgery. Influence of previous abdominal surgery on surgical outcomes between laparoscopic and open surgery in elderly patients with colorectal cancer: subanalysis of a large multicenter study in Japan. J Gastroenterol. 2017 Jun;52(6):695-704. doi: 10.1007/s00535-016-1262-5. Epub 2016 Sep 20. PMID 27650199
- [Result] Nakamura T, Sato T, Naito M, Ogura N, Yamanashi T, Miura H, Tsutsui A, Yamashita K, Watanabe M. Laparoscopic Surgery is Useful for Preventing Recurrence of Small Bowel Obstruction After Surgery for Postoperative Small Bowel Obstruction. Surg Laparosc Endosc Percutan Tech. 2016 Feb;26(1):e1-4. doi: 10.1097/SLE.0000000000000238. PMID 26771166